CLINICAL TRIAL: NCT02601300
Title: A Phase 2, Open-Label, Multicenter Study to Explore the Efficacy and Safety of MONGERSON (GED-0301) in Subjects With Active Ulcerative Colitis.
Brief Title: An Efficacy and Safety Study of Mongersen (GED-0301) in Subjects With Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GED-0301-UC-002
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis; GED-0301; Mongersen; Efficacy; Safety
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GED0301

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GED-0301 160 mg once daily (QD) (Experimental): Patients will receive oral GED-0301 160 mg once daily (QD)for duration of 52 week treatment.
  Interventions: Drug: GED-0301

INTERVENTIONS:
Drug: GED-0301
  Other Names: Mongersen

SUMMARY:
This is a phase 2, open-label, multicenter study to explore the efficacy and safety of oral GED- 0301 in subjects with active UC, defined as a modified Mayo score (MMS) ≥ 4 and ≤ 9 and a Mayo endoscopic subscore≥ 2.

Approximately 40 subjects will be enrolled using an Interactive Voice Response System (IVRS) or an Interactive Web Response System (IWRS) to receive open-label, oral GED-0301 160 mg for duration of 52 week treatment. Enrollment of subjects with previous exposure to TNF-α blockers will be limited to approximately 15 subjects. The number of subjects with extensive colitis is targeted to comprise approximately 50% of the entire study population.

DETAILED DESCRIPTION:
Eligible subjects will have the Baseline Visit (Week 0/ Visit 2) and receive the following treatments:

* Induction Phase - GED-0301 160 mg once daily (QD) for 8 weeks;
* Extension Phase - GED-0301 160 mg on alternating dosing schedule (GED-0301 160 mg QD for 4 weeks, followed by 4 weeks without GED-0301 treatment) for an additional 44 weeks. Subjects who do not achieve at least a 20% decrease in partial mayo score (PMS) from baseline at Week 12 will be discontinued from the study.

Clinical, safety, and pharmacokinetic (PK) data will be evaluated on an ongoing basis, however, if the response to treatment is lower than expected (eg, ≤2 subjects achieving clinical remission based on modified Mayo score (MMS)) when 50% of the subjects complete Week 8, or discontinue before Week 8, the study team will review available data (clinical, safety, and PK) to evaluate if the study conduct should be modified.

This evaluation will be based on clinical judgment and the following guidance

* Consider starting a new cohort of subjects using a QD dose up to 320 mg if there is endoscopic or histologic evidence of proximal colon benefit but limited or no distal colon drug exposure/efficacy. Also, there is evidence of potential overall efficacy (total Mayo score (TMS), MMS,PMS) outcomes and acceptable safety (adverse events (AEs)/vitals/clinical laboratory test results) and exposure (PK).
* Consider to terminate the study if there is no evidence of drug exposure/efficacy in the colon observed by endoscopy or biopsy nor evidence of potential overall efficacy (TMS, MMS, PMS) outcomes or unacceptable safety(AEs/labs/vitals) or exposure (PK).
* Continue the study with the GED-0301 160 mg QD dose. If the GED-0301 160 mg QD dose group is discontinued and a new dose group is added, an additional 40 subjects will be enrolled in the new dose group. Subjects enrolled subsequent to the decision to adjust the dose of GED-0301, will receive the following treatments:
* Induction Phase - GED-0301, up to 320 mg QD, for 8 weeks;
* Extension Phase- GED-0301, up to 320 mg on alternating dosing schedule (GED-0301, up to 320 mg QD for 4 weeks, followed by 4 weeks without GED-0301 treatment) for an additional 44 weeks. Subjects who do not achieve at least a 20% decrease in the PMS from baseline at Week 12 will be discontinued from the study. Actively enrolled subjects will not be affected by the dose adjustment. Subjects receiving corticosteroids at baseline will start tapering their corticosteroids at Week 8 (the end of the Induction Phase) if they achieve clinical response, defined as a decrease from baseline of at least 2 points and at least 25%, along with a reduction in the RBS of at least 1 point or an absolute RBS ≤ 1 in the MMS. The endoscopy subscore assessed by the investigator will be used for the calculation of the Week 8 MMS.

The study will consist of 4 phases:

* Screening Phase - up to 4 weeks
* Induction Phase - 8 weeks
* Extension Phase - 44 weeks
* Observational Follow-up Phase - 4 weeks Subjects who complete the Extension Phase, and those subjects who prematurely discontinue from the study for any reason, will enter the post-treatment Observational Follow-up Phase, the 4-week period after the last dose of Investigational Product(IP). The study will be conducted in compliance with International Conference on Harmonisation (ICH) Good Clinical Practices (GCPs).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
  2. Subject is able to understand and voluntarily sign an informed consent form (ICF)prior to conducting any study related assessments/procedures.
  3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
  4. Subject must have diagnosis of Ulcerative Colitis (UC) with a duration of at least 3 months prior to screening.
  5. Subject must have moderate to severe Ulcerative Colitis (UC), defined as Modified Mayo score (MMS) ≥ 4 to ≤ 9 with rectal bleeding subscore (RBS) ≥ 1 at screening.
  6. Subject must have a Mayo endoscopic subscore ≥ 2 at screening.
  7. Subject must have failed or experienced intolerance to at least one of the following:

     aminosalicylates; budesonide; systemic corticosteroids; immunosuppressants (eg,6-mercaptopurine (6-MP), or azathioprine (AZA)) or Tumor necrosis factor (TNF)-α blockers (eg, infliximab, adalimumab, or golimumab)
  8. Subject must meet the following laboratory criteria:

     1. White blood cell count ≥ 3000/mm3 (≥ 3.0 X 109/L)
     2. Platelet count ≥ 100,000/mm3 (≥ 100 X 109/L)
     3. Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
     4. Aspartate transaminase (AST/serum glutamic oxaloacetic transaminase (SGOT)) and alanine transaminase (ALT/serum pyruvic transaminase (SGPT)2.5 X upper limit of normal (ULN)
     5. Total bilirubin ≤ 2 mg/dL (≤ 34 μmol/L) unless there is a confirmed diagnosis of Gilbert's disease
     6. Hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L)
     7. Activated partial thromboplastin time (APTT) 1.5 X ULN
  9. Females of childbearing potential (FCBP) must have a negative pregnancy test at the Screening and Baseline Visits. While on Investigational Product (IP)and for at least 28 days after taking the last dose of Investigational Product (IP), females of childbearing potential (FCBP) who engage in activity in which conception is possible must use one of the approved contraceptive options described below: Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom PLUS 1 additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
  10. Male subjects (including those who have had a vasectomy) when engaging in sexual activity with females who are able to become pregnant must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on Investigational Product (IP) and for at least 28 days after the last dose.

      Exclusion Criteria:
* The presence of any of the following will exclude a subject from enrollment:

  1. Subject has a diagnosis of Crohn's Disease (CD), indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis.
  2. Subject has ulcerative colitis restricted to distal 15 cm or less (eg, ulcerative proctitis).
  3. Subject had surgery as a treatment for ulcerative colitis (UC)or who, in the opinion of the Investigator, is likely to require surgery for ulcerative colitis (UC) during the study.
  4. Subject has clinical signs suggestive of fulminant colitis or toxic megacolon.
  5. Subject is stool positive for any enteric pathogen or Clostridium difficile (C. difficile) toxin at screening.
  6. Subject has history of colorectal cancer or colorectal dysplasia.
  7. Prior treatment with more than 2 Tumor necrosis factor (TNF)-α blockers (eg, infliximab, adalimumab, or golimumab).
  8. Prior treatment with any integrin antagonists (eg, natalizumab or vedolizumab).
  9. Use of Tumor necrosis factor (TNF)-α blockers within 8 weeks of the screening.
  10. Subject had prior treatment with mycophenolic acid, tacrolimus, sirolimus, cyclosporine, thalidomide or apheresis (eg, Adacolumn®) for the treatment of ulcerative colitis (UC). In addition, prior use of any of these treatment modalities for an indication other than ulcerative colitis (UC) within 8 weeks of screening is also excluded.
  11. Subject has received intravenous (IV) corticosteroids within 2 weeks of screening.
  12. Subject has received topical treatment with 5 aminosalicylic acid (5-ASA) or corticosteroid enemas or suppositories within 2 weeks of screening.
  13. Subject has received total parenteral nutrition (TPN) within 4 weeks of screening.
  14. Subject has a history of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the investigator's opinion, would prevent the subject from participation in the study.
  15. Subject has any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she was to participate in the study or confounds the ability to interpret data from the study.
  16. Subject is pregnant or breastfeeding.
  17. Subject has a history of any of the following cardiac conditions within 6 months of screening: myocardial infarction, acute coronary syndrome, unstable angina, new onset atrial fibrillation, new onset atrial flutter, second- or third-degree atrioventricular block, ventricular fibrillation, ventricular tachycardia, heart failure, cardiac surgery, interventional cardiac catheterization (with or without a stent placement), interventional electrophysiology procedure, or presence of implanted defibrillator.
  18. Subject has a known active current or history of medically important recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease and Herpes zoster), human immunodeficiency virus (HIV), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) or oral antibiotics within 4 weeks of screening.
  19. Subject has a history of congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease).
  20. Subject has a history of malignancy, except for:

      1. Treated (ie, cured) basal cell or squamous cell in situ skin carcinomas
      2. Treated (ie, cured) cervical intraepithelial neoplasia or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years
  21. Subject has received investigational drug or device within 1 month of screening.
  22. Subject has a history of alcohol, drug, or chemical abuse within the 6 months prior to screening.
  23. Subject has a known hypersensitivity to oligonucleotides or any ingredient in the Investigational Product (IP).
  24. Subject has prior treatment with GED-0301 or participated in a clinical study involving GED-0301.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Usiskin, M.D, Study Director — Celgene Corporation
Locations (36):
- United States (20):
  - Macks Research Group, Newport Beach, California
  - Medical Associates Research Associates, San Diego, California
  - Florida Research Network, LLC, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - University of Kentucky, Lexington, Kentucky
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Concorde Medical Group, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Gastroenterology Center of The Midsouth PC, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Dean Medical Center, Madison, Wisconsin
- Bulgaria (3):
  - Multiprofile Hospotal for Active Treatment- Sveti Nikolay Chudotvoretz - LOM EOOD, Lom
  - Multiprofile Hospital for Active Treatment Doverie AD, Sofia
  - Multiprofile Hospital for Active Treatment Sveti Panteleimon - Sofia AD, Sofia
- Canada (3):
  - GI Research Institute, Vancouver, British Columbia
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
- Pandy Kalman Megyei Korhaz, Siófok, Hungary
- Poland (4):
  - Centrum Medyczne sw. Lukasza, Częstochowa
  - Endoskopia Sp. z o.o., Sopot
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - IBD Centrum s.r.o., Bratislava
  - KM Management, spol. s r.o., Nitra
  - GASTRO I., s.r.o., Prešov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 21 study centers within the United States, Bulgaria, Poland, Slovakia and Canada.
Pre-assignment Details: Participants were 18 years of age and older with active ulcerative colitis for 3 months prior to screening, had a modified Mayo score (MMS) ≥ 4 to ≤ 9 absolute rectal bleeding (RBS) subscore ≥ 1 at screening, a mayo endoscopic subscore ≥ 2 at screening and must have had a therapeutic failure or been intolerant to other therapies.
Groups:
- Mongersen (Weeks 0-52): Participants received oral mongersen 160 mg tablets daily for 8 weeks during the induction phase, followed by 160 mg tablets daily on an alternating dosing schedule for 4 weeks, followed by a 4 week break, (4 weeks on investigational product (IP), followed by 4 weeks off) for an additional 44 weeks during the extension phase, weeks 8 through 52). Participants who did not achieve at least a 20% decrease in a partial Mayo score (PMS) from baseline at Week 12 were discontinued from the study.
Period: Induction Phase
Arm/Group | Mongersen (Weeks 0-52)
Started | 41
Completed | 38
Not Completed | 3
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1
Period: Extension Phase
Arm/Group | Mongersen (Weeks 0-52)
Started | 35 (3 completed induction phase; did not enter extension due to withdrawal and lack of efficacy)
Treated With IP | 34
Completed | 18
Not Completed | 17
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population includes all participants who received at least 1 dose of investigational product.
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 2
  White | 37
  Other | 1
Duration of Ulcerative Colitis [Mean (Standard Deviation); unit: years] | 9.91 (9.107)
Baseline Modified Mayo Score (MMS) [Mean (Standard Deviation); unit: units on a scale] — A modification to the total Mayo score (TMS) was implemented. The MMS was based on the stool frequency, rectal bleeding and endoscopy subscores of the total Mayo score, and excluded the Physician's Global subscore, since this was a global measure that is subjective in nature. The MMS ranges from 0 to 9 points, with higher scores indicating greater disease severity.
  units on a scale | 6.5 (1.50)
Baseline Mayo Endoscopic Subscore [Mean (Standard Deviation); unit: units on a scale] — The Mayo endoscopic subscore is one of the components of the Mayo score and ranges from 0 - 3 points and is defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration)
  units on a scale | 2.6 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission in the Modified Mayo Score (MMS) at Week 8
Description: Clinical remission was defined as a modified Mayo score of ≤ 2, with no individual subscore > 1, at Week 8. The MMS was based on a modification of the total Mayo score (TMS) which included the stool frequency, rectal bleeding, and endoscopic subscores of the TMS and excluded the Physician's Global Assessment (PGA) subscore, since this was a global measure that is subjective in nature. The MMS ranges from 0 to 9 points with higher scores indicating greater disease severity. The endoscopy subscores was centrally reviewed. Two-sided confidence intervals for the within-group percentage were based on the Wilson score method.
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handing missing data was non-responder imputation (NRI) method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for clinical remission.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 17.1 [8.5 to 31.3]

2. Secondary Outcome: Percentage of Participants Who Achieved a Modified Mayo Score of ≤ 2, With Rectal Bleeding Subscore (RBS) of 0 and Stool Frequency Subscore (SFS) and Mayo Endoscopic Subscore ≤ 1 at Week 8
Description: A MMS was used to evaluate disease activity using 3 components: stool frequency, rectal bleeding and endoscopy; the MMS ranges from 0-9 with higher scores indicating greater disease severity.
  Stool frequency subscore was defined as 0-3:
  0 = Normal number of stools for patient
  1. = 1-2 stools per day more than normal
  2. = 3-4 stools more than normal
  3. = 5 or more stools more than normal
  Rectal bleeding (subscore 0-3) was defined as:
  0 = No blood seen
  1. = Streaks of blood with stool less than half the time
  2. = Obvious blood with stool most of the time
  3. = Blood alone passes
  Endoscopic subscore: Findings were defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration)
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handling missing data was NRI method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for the MMS response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 14.6 [6.9 to 28.4]

3. Secondary Outcome: Percentage of Participants Who Achieved a Mayo Endoscopic Subscore of ≤ 1 at Week 8
Description: A Mayo endoscopic subscore of ≤ 1 was assessed and evaluated in participants who achieved a Mayo endoscopic subscore at Week 8. The endoscopy subscore findings are defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration) The endoscopy scores were centrally reviewed. Two-sided 95% CIs for the within-group percentage were based on the Wilson score method.
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handling missing data was NRI method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for Mayo Endoscopic Subscore.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 19.5 [10.2 to 34.0]

4. Secondary Outcome: Percentage of Participants Who Achieved a Mayo Endoscopic Subscore of ≤ 1 by Individual Segment at Week 8
Description: A Mayo endoscopic subscore by individual segment (rectum, sigmoid, descending colon, transverse colon, ascending colon/cecum) of ≤ 1 was evaluated at week 8.
  The endoscopy subscore findings are defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration) The endoscopy scores were centrally reviewed. Two-sided 95% CIs for the within-group percentage were based on the Wilson score method.
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. Only participants with sufficient data for response determination in each segment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants
  Rectum: number analyzed (Participants) | 37
  Rectum | 27.0 [15.4 to 43.0]
  Sigmoid: number analyzed (Participants) | 37
  Sigmoid | 27.0 [15.4 to 43.0]
  Descending Colon: number analyzed (Participants) | 35
  Descending Colon | 54.3 [38.2 to 69.5]
  Transverse Colon: number analyzed (Participants) | 28
  Transverse Colon | 60.7 [42.4 to 76.4]
  Ascending Colon/Cecum: number analyzed (Participants) | 25
  Ascending Colon/Cecum | 80.0 [60.9 to 91.1]

5. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Modified Mayo Score at Week 8
Description: Clinical response in the MMS was defined as a decrease from baseline in the MMS of at least 2 points and at least 25%, along with a reduction in the RBS of at least 1 point or an absolute RBS ≤ 1. The MMS was based on the stool frequency, rectal bleeding, and endoscopic subscores of the TMS and excluded the PGA subscore. The MMS ranges from 0 to 9 points with higher scores indicating greater disease severity. The RBS was defined as:
  0 = No blood seen
  1. = Streaks of blood with stool less than half the time
  2. = Obvious blood with stool most of the time
  3. = Blood alone passes The daily bleeding score represents the most severe bleeding score represents the most severe bleeding of the day.
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handling missing data was NRI method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for MMS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 36.6 [23.6 to 51.9]

6. Secondary Outcome: Percentage of Participants Who Achieved a Mayo Endoscopic Response at Week 8
Description: Endoscopic response was defined as a decrease from baseline of at least 1 point in the Mayo endoscopic subscore. The Mayo endoscopy subscore findings are defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration) The endoscopy subscores were centrally reviewed. Two-sided 95% CIs for the within-group percentage were based on the Wilson score method.
Time Frame: Baseline and Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handling missing data was NRI method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for Mayo endoscopic response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 31.7 [19.6 to 47.0]

7. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Remission in the Total Mayo Score (TMS) at Week 8
Description: Clinical remission in total Mayo score was defined as a total Mayo score of ≤ 2, with no individual subscore >1. The TMS is an instrument designed to measure disease activity of ulcerative colitis. The TMS ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease.
  * Stool frequency subscore (SFS)
  * Rectal bleeding subscore (RBS)
  * Endoscopic subscore
  * Physician's Global Assessment (PGA)
Time Frame: Baseline to Week 8
Population: The intent to treat population included all participants who received at least one dose of IP. The primary approach to handling missing data was NRI method, where participants who had insufficient data for response determination at Week 8 were considered non-responders for Total Mayo score.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 9.8 [3.9 to 22.5]

8. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Total Mayo Score at Week 8
Description: Clinical response in the TMS was defined as a decrease from baseline in the TMS of ≥ 3 points and ≥ 30%, along with a reduction in the RBS of ≥ 1 point or an absolute RBS of ≤ 1 at Week 8. The TMS is an instrument designed to measure disease activity of ulcerative colitis. The TMS ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease.
  * Stool frequency subscore
  * Rectal bleeding subscore
  * Endoscopic subscore
  * Physician's Global Assessment
Time Frame: Baseline to Week 8
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mongersen (Weeks 0-52)
Number analyzed (Participants) | 41
percentage of participants | 36.6 [23.6 to 51.6]

9. Secondary Outcome: The Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as any adverse event (AE) occurring or worsening on or after the first treatment of mongersen and up to 28 days after the last mongersen dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale: Mild = asymptomatic or mild symptoms; clinical or diagnostic observations only; Moderate = Symptoms cause moderate discomfort; Severe (could be non-serious or serious) = symptoms causing severe discomfort/pain.
Time Frame: From the first day of mongersen until 28 days after the last dose of IP or at follow-up visit, whichever occurred earlier; maximum duration of treatment was 56 weeks
Population: Safety population included all participants who were enrolled and received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Groups:
- Mongersen Total Mongersen Exposure Period: Participants who received oral mongersen 160 mg tablets during the induction phase and the extension phase, with dosing starting on the first mongersen dose of the induction phase and ended at the last follow-up date up to 28 days after the last mongersen dose (either in the induction or the extension phase)
Arm/Group | Mongersen Total Mongersen Exposure Period
Number analyzed (Participants) | 41
Participants
  Any TEAE | 30
  Any IP-Related TEAE | 6
  Any Severe TEAE | 5
  Any Serious TEAE (SAE) | 5
  Any Serious IP-Related TEAE | 0
  Any TEAE Leading to IP Withdrawal | 4
  Any TEAE Leading to IP Interruption | 1
  Any TEAE Leading to Death | 0

ADVERSE EVENTS:
Time Frame: From the first day of mongersen until 28 days after the last dose of IP or at follow-up visit, whichever occurred earlier; the maximum duration of treatment was 56 weeks
Groups:
- Mongersen (Induction Phase: Weeks 0-8): Participants received oral mongersen 160 mg tablets daily for 8 weeks during the induction phase.
- Mongersen (Extension Phase: Weeks 8-52): Participants received oral mongersen 160 mg tablets daily on an alternating dosing schedule for 4 weeks, followed by a 4 week break, (4 weeks on investigational product (IP), followed by 4 weeks off) for an additional 44 weeks during the extension phase. Participants who did not achieve at least a 20% decrease in a partial Mayo score (PMS) from baseline at Week 12 were discontinued from the study.
Arm/Group | Mongersen (Induction Phase: Weeks 0-8) | Mongersen (Extension Phase: Weeks 8-52)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/41 | 4/34
Other Adverse Events (participants affected / at risk) | 0/41 | 14/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mongersen (Induction Phase: Weeks 0-8) (N=41) | Mongersen (Extension Phase: Weeks 8-52) (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mongersen (Induction Phase: Weeks 0-8) (N=41) | Mongersen (Extension Phase: Weeks 8-52) (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission and defer publication to permit patent applications.